CLINICAL TRIAL: NCT00721552
Title: Sitagliptin Prophylaxis for Glucocorticoid-Induced Impairment of Glucose Metabolism and Beta-Cell Dysfunction in Males With the Metabolic Syndrome X: A Randomized, Placebo-controlled, Double-blind Intervention Study With a 2x2 Factorial Design
Brief Title: Sitagliptin Prophylaxis for Glucocorticoid-Induced Impairment of Glucose Metabolism in Males With the Metabolic Syndrome
Acronym: SPHINX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M. Diamant, Prof. M. Diamant, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: DC2008Pred002; Eudract 2008-004985-25
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus; Steroid Diabetes; Glucocorticoid-induced Diabetes; Beta-cell Function
Keywords: beta-cell function; glucocorticoid-induced diabetes; glucocorticoid; DPP-4 inhibitors; sitagliptin; diabetes mellitus; steroid diabetes; insulin resistance; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Sitagliptin Phosphate; Prednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- I (Experimental): prednisolone + sitagliptin
  Interventions: Drug: Sitagliptin 100 mg; Drug: Prednisolone 30 mg
- II (Experimental): prednisolone + sitagliptin-placebo
  Interventions: Drug: Prednisolone 30 mg; Drug: Sitagliptin-placebo
- III (Experimental): prednisolone-placebo + sitagliptin
  Interventions: Drug: Sitagliptin 100 mg; Drug: Prednisolone-placebo
- IV (Placebo Comparator): prednisolone-placebo + sitagliptin-placebo
  Interventions: Drug: Sitagliptin-placebo; Drug: Prednisolone-placebo
- Healthy controls (No Intervention): 12 healthy men will be included to assess postprandial microvascular function.
- Type 2 diabetic subjects (No Intervention): 12 men with type 2 diabetes will be included in order to assess postprandial microvascular function.

INTERVENTIONS:
Drug: Sitagliptin 100 mg — 28 days administration of 100 mg daily
  Other Names: Januvia; MK-0431; ATC A10BH01
  Arms: I; III
Drug: Prednisolone 30 mg — 14 days administration of 30 mg daily
  Other Names: prednison; ATC H02AB06
  Arms: I; II
Drug: Sitagliptin-placebo — 28 days administration once daily
  Arms: II; IV
Drug: Prednisolone-placebo — 14 days administration once daily
  Arms: III; IV

SUMMARY:
The investigators will assess whether the DPP-inhibitor sitagliptin will ameliorate glucocorticoid-induced impairment of glucose metabolism and beta-cell dysfunction and thus could be used as a prophylaxis for glucocorticoid-induced diabetes. Therefore the investigators will administer in males with the metabolic syndrome 30 mg prednisolone daily for two weeks and give simultaneously sitagliptin 100 mg daily. Subjects will undergo at baseline and after two weeks of treatment several tests to assess changes in glucose metabolism.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, placebo-controlled, double-blind, 2x2 factorial-designed intervention trial. The pharmacological intervention for prednisolone/prednisolone-placebo is 14 days and for sitagliptin/sitagliptin-placebo 28 days. Subjects fulfilling the IDF criteria26 for the metabolic syndrome (aged 35-65; n=60) will be randomized to one of four groups: I) prednisolone 30 mg and sitagliptin 100 mg daily; II) prednisolone 30 mg and sitagliptin-placebo daily; III) prednisolone-placebo and sitagliptin 100 mg daily; IV) prednisolone-placebo and sitagliptin-placebo daily. Before and at day 14 of treatment subjects will undergo a standardized mixed-meal test in order to assess glucose disposal and beta-cell function (by modeling analysis). During these meal tests, plasma concentrations of (total and active) GLP-1, GIP, glucagon and additional biomarkers will be assessed. A combined hyperglycemic-euglycemic clamp will be performed at baseline and at day 13 of treatment to assess insulin sensitivity and insulin secretion. During the euglycemic clamp adipose tissue and muscle biopsies will be obtained, both in fasting and under hyperinsulinemic conditions. At baseline and at day 28 of treatment, a 7-point OGTT will be performed to assess time to restoration of glycemic control. Body composition, body fat distribution and liver fat content, measured by respectively bio-impedance analysis and magnetic resonance imaging/spectroscopy (MRI/MRS), will be assessed at baseline and after 28 days of treatment. Blood pressure will be assessed at baseline and after two weeks of treatment. Microvascular function will be assessed with capillary videomicroscopy both at baseline and after two weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males
* Modified from IDF criteria for the metabolic syndrome:

  * Waist circumference ≥ 94 cm
* And at least 2 or more of the following criteria:

  * TG ≥ 1.7 mmol/L
  * HDL cholesterol < 1.03 mmol/L
  * Blood pressure >130/85 mmHg (average of three measurements) or treatment of previously diagnosed hypertension
  * Fasting plasma glucose level (FPG) ≥ 5.6 mmol/L (but no diabetes)

Exclusion Criteria:

* An allergic or anaphylactic reaction to prednisolone treatment in the past
* Clinically relevant history or presence of any medical disorder, which are mentioned in the Summary of Product Characteristics (SPC) as contraindication for the use of prednisolone
* Glucocorticosteroid use during the last three months prior to the first dose
* Participation in an investigational drug trial within 90 days prior to the first dose
* Donation of blood ( > 100 mL) within 90 days prior to the first dose
* History of or current abuse of drugs or alcohol (>14 U/week)
* Use of grapefruit products during the study period
* Recent changes in weight and/or physical activity
* Serious mental impairment or language problems i.e. preventing to understand the study protocol/aim
* Diabetes mellitus (defined as FPG ≥ 7.0 mmol/l and/or 2hPG ≥ 11.1 mmol/l)
* Serious pulmonary, cardiovascular, hepatic (ALT, AST more than 3x ULN) or renal disease (serum creatinine > 135 micromol/L)
* History of cardiovascular disease, such as myocardial infarction, cerebrovascular accident.
* Major psychiatric disorder, depression
* All diseases that induce changes in the hypothalamic-pituitary-adrenal (HPA) axis
* Malignant disease
* All other relevant medical disorders that potentially interfere with this trial.
* All medication interfering with study drug or interfering with study endpoints/hypotheses

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance as assessed by the area under the curve for glucose (AUCgluc) during a standardized meal test. | 14 days

SECONDARY OUTCOMES:
Incretin secretion during standardized meal test | 14 days
Insulin sensitivity | 14 days
Microvascular function: fasting and postprandial | 14 days
Body composition, body fat distribution and intra organ fat accumulation | 28 days
Molecular mechanisms in subcutaneous adipose tissue | 14 days
Blood pressure and hemodynamic parameters | 28 days
Biomarkers such as lipoproteins, adipocytokines, and markers of systemic inflammation | 14 days
Time to recovery after cessation of the two-week prednisolone treatment | 28 days
Beta-cell function as determined by hyperglycemic clamp tests and modeling analysis from mixed-meal tests. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Diamant, Md PhD, Principal Investigator — VUmc Diabetes Center, Amsterdam, The Netherlands
Locations (1):
- VUmc Diabetes Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Genugten RE, van Raalte DH, Muskiet MH, Heymans MW, Pouwels PJ, Ouwens DM, Mari A, Diamant M. Does dipeptidyl peptidase-4 inhibition prevent the diabetogenic effects of glucocorticoids in men with the metabolic syndrome? A randomized controlled trial. Eur J Endocrinol. 2014 Feb 4;170(3):429-39. doi: 10.1530/EJE-13-0610. Print 2014 Mar. PMID 24297090
- [Derived] van Genugten RE, Serne EH, Heymans MW, van Raalte DH, Diamant M. Postprandial microvascular function deteriorates in parallel with gradual worsening of insulin sensitivity and glucose tolerance in men with the metabolic syndrome or type 2 diabetes. Diabetologia. 2013 Mar;56(3):583-7. doi: 10.1007/s00125-012-2783-y. Epub 2012 Nov 24. PMID 23178932